CLINICAL TRIAL: NCT02430376
Title: dbGaP Protocol: Genetic Variants Associated With Pentalogy of Cantrell
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915111; 15-H-N111
Record Dates: First submitted 2015-04-25; First posted 2015-04-30 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03-07

CONDITIONS: Pentalogy of Cantrell
Keywords: Non-Muscle Myosin
MeSH Terms: conditions — Pentalogy of Cantrell

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective

SUMMARY:
Background:

Pentalogy of Cantrell (POC) is a syndrome that involves many heart abnormalities as well as large defects in the chest and abdominal wall. This often results in the heart and other organs being present outside the body at birth. Surgeons have learned to replace them and repair the heart. Researchers want to find possible gene changes that cause POC. To do this, they want to study data from the Pediatric Cardiovascular Genetics Consortium (PCGC) Cohort. The PCGC collects data and DNA samples from people with heart diseases and their families

Objectives:

- To find gene mutations in people with Pentalogy of Cantrell (POC) or other related syndromes.

Eligibility:

- PCGC data and DNA samples that are open to study by the public.

Design:

* Researchers will study the data from the PCGC.
* The gene testing being done in this study was consented to in the original studies. No new consent or waiver request is required.
* The study will last 1 year.

DETAILED DESCRIPTION:
The purpose of this protocol is to identify genetic mutations in patients with the diagnosis of Pentalogy of Cantrell (POC) or other related syndromes. We will be looking for any exomic/genomic mutations that could be associated with this syndrome. We have produced a mouse model with a mutation in the gene encoding nonmuscle myosin IIB which exhibit problems with ventral wall closure, including extrathoracic location of the heart (ectopia cordis) and defects in the abdominal wall with protrusion of the guts and liver. These mice have severe defects in both the heart and brain, and resemble humans born with POC, who manifest these same abnormalities, and so we take a special interest in mutations in nonmuscle myosin proteins.

ELIGIBILITY:
* We will analyze data from subjects from congenital cardiovascular disease databases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3280 (Actual)
Dates: Start 2015-04-25; Primary Completion 2016-03-23 (Actual); Study Completion 2016-03-23 (Actual)

PRIMARY OUTCOMES:
To identify novel genetic mutations associated with the disease Pentalogy of Cantrell | Ongoing

SECONDARY OUTCOMES:
To identify the molecular mechanisms underlying the congenital disease Pentalogy of Cantrell, to aid in the development of novel therapeutic strategies. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Adelstein, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States